CLINICAL TRIAL: NCT02201316
Title: An Open-label, Randomised, Single Dose, Three-Way Crossover, Six Sequence, Pilot Study to Determine the Relative Bioavailability of Mosapride 5mg From Two Candidate Formulations of GR107719B Relative to One 5mg Tablet of Reference Mosapride Citrate (Gasmotin) in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: A Pilot Study to Determine the Relative Bioavailability of Mosapride 5mg From Two Candidate Formulations of GR107719B Relative to One 5mg Tablet of Reference Mosapride Citrate (GASMOTIN™) in Healthy Adult Human Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200940
Record Dates: First submitted 2013-12-19; First posted 2014-07-28 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Gastritis
Keywords: Healthy adult human subjects; Mosapride citrate anhydrous; Bioequivalence; Dyspepsia
MeSH Terms: conditions — Gastritis; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (ABC) (Experimental): Subjects will receive treatments in the sequence ACB where, A=Single dose of reference mosapride citrate 5mg (GASMOTIN); B= Single dose of formulation 1 GR107719B 5mg (mosapride citrate); C= Single dose of formulation 2 GR107719B 5mg (mosapride citrate). All treatments will be administered orally in fasted state. Each treatment will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Reference mosapride citrate (GASMOTIN); Drug: GR107719B (Formulation 1); Drug: GR107719B (Formulation 2)
- Sequence 2 (ACB) (Experimental): Subjects will receive treatments in the sequence ACB where, A=Single dose of reference mosapride citrate 5mg (GASMOTIN); B= Single dose of formulation 1 GR107719B 5mg (mosapride citrate); C= Single dose of formulation 2 GR107719B 5mg (mosapride citrate). All treatments will be administered orally in fasted state. Each treatment will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Reference mosapride citrate (GASMOTIN); Drug: GR107719B (Formulation 1); Drug: GR107719B (Formulation 2)
- Sequence 3 (BAC) (Experimental): Subjects will receive treatments in the sequence BAC where, A=Single dose of reference mosapride citrate 5mg (GASMOTIN); B= Single dose of formulation 1 GR107719B 5mg (mosapride citrate); C= Single dose of formulation 2 GR107719B 5mg (mosapride citrate). All treatments will be administered orally in fasted state. Each treatment will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Reference mosapride citrate (GASMOTIN); Drug: GR107719B (Formulation 1); Drug: GR107719B (Formulation 2)
- Sequence 4 (BCA) (Experimental): Subjects will receive treatments in the sequence BCA where, A=Single dose of reference mosapride citrate 5mg (GASMOTIN); B= Single dose of formulation 1 GR107719B 5mg (mosapride citrate); C= Single dose of formulation 2 GR107719B 5mg (mosapride citrate). All treatments will be administered orally in fasted state. Each treatment will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Reference mosapride citrate (GASMOTIN); Drug: GR107719B (Formulation 1); Drug: GR107719B (Formulation 2)
- Sequence 5 (CAB) (Experimental): Subjects will receive treatments in the sequence CAB where, A=Single dose of reference mosapride citrate 5mg (GASMOTIN); B= Single dose of formulation 1 GR107719B 5mg (mosapride citrate); C= Single dose of formulation 2 GR107719B 5mg (mosapride citrate). All treatments will be administered orally in fasted state. Each treatment will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Reference mosapride citrate (GASMOTIN); Drug: GR107719B (Formulation 1); Drug: GR107719B (Formulation 2)
- Sequence 6 (CBA) (Experimental): Subjects will receive treatments in the sequence CBA where, A=Single dose of reference mosapride citrate 5mg (GASMOTIN); B= Single dose of formulation 1 GR107719B 5mg (mosapride citrate); C= Single dose of formulation 2 GR107719B 5mg (mosapride citrate). All treatments will be administered orally in fasted state. Each treatment will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Reference mosapride citrate (GASMOTIN); Drug: GR107719B (Formulation 1); Drug: GR107719B (Formulation 2)

INTERVENTIONS:
Drug: Reference mosapride citrate (GASMOTIN) — Reference mosapride citrate (GASMOTIN) 5mg will be supplied as caplet shaped tablet embossed with P218 and film-coated; administer orally with approximately 240 mL of water.
Drug: GR107719B (Formulation 1) — GR107719B (Formulation 1) 5 mg will be supplied as L-HPC disintegrant caplet shaped tablet, embossed and film-coated; administer orally with approximately 240 mL of water.
Drug: GR107719B (Formulation 2) — GR107719B (Formulation 2) 5 mg will be supplied as caplet shaped tablet, embossed and film-coated; administer orally with approximately 240 mL of water.

SUMMARY:
This study aims to determine the relative bioavailability of two candidate formulations of mosapride citrate 5mg tablets compared the reference product GASMOTIN (mosapride citrate 5mg) from Dainippon Pharmaceutical Company in healthy adult subjects. This will be an open-label, randomised, single dose, three-way crossover, six sequence study. Subjects will receive a single oral dose separated by at least 7 days and no greater than 14 days washout period. This study is required to select a candidate mosapride citrate (GR107719B) formulation for further development and provide data to allow the design of a future pivotal bioequivalence study. The candidate formulations will be compared with the innovator GASMOTIN. GASMOTIN is a trademark of Dainippon Sumitomo Pharmaceutical Company.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) and body mass index within the range 19 - 24.9 kg/m^2 (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (MlU/mL) and estradiol < 40 picograms per mililiter (pg/mL) [<147 picomole per liter] is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotrophin (hCG) test at screening or prior to dosing AND; Agrees to use one of the contraception methods listed in protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up contact visit; OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up contact visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase, alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiograms obtained over a brief recording period: QTcF < 450 msec

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (100 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational product.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2014-03-18 (Actual); Study Completion 2014-03-18 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics (PK) parameters of mosapride following administration of two candidate tablet formulations of mosapride citrate (GR107719B) relative to reference mosapride citrate (GASMOTIN) | Day 1 of each treatrment period (Pre dose and 0.25 hour (h), 0.5 h, 0.75 h, 1 h, 1.33 h, 1.67 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h post dose)
  PK parameters include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)] and area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration [AUC(0-t)]

SECONDARY OUTCOMES:
PK parameters of two candidate tablet formulations of mosapride citrate (GR107719B) relative to reference mosapride citrate tablets (GASMOTIN) | Day 1 of each treatrment period (Pre dose and 0.25 hour (h), 0.5 h, 0.75 h, 1 h, 1.33 h, 1.67 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h post dose)
  PK parameters include: Percentage of AUC (0-∞) obtained by extrapolation (%AUCex) time of occurrence of Cmax (tmax), terminal phase half-life (t1/2).
Safety and tolerability assessment as assessed by review of adverse events (AEs) | Up to 51 days
Safety and tolerability assessment as assessed by vital signs | Up to 51 days
  Vital sign measurements will include systolic and diastolic blood pressure, and pulse rate.
Safety and tolerability assessment as assessed by clinical laboratory values | Up to 51 days
  Clinical laboratory assessments will include hematology, clinical chemistry, routine urinalysis and additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India

REFERENCES:
- See also: Results for study 200940 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200940?search=study&search_terms=200940#rs